CLINICAL TRIAL: NCT01273831
Title: Study of Effects of Cisatracurium and Atracurium on Intraocular Pressure
Brief Title: Effect of Cisatracurium Versus Atracurium on Intraocular Pressure in Patients Underwent General Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy/Associate Professor of Medical Education, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: ASD-1213-10
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2009-07

CONDITIONS: Intraocular Pressure
Keywords: intraocular pressure, anesthesia,cisatracurium,atracurium.
MeSH Terms: interventions — Atracurium; cisatracurium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- atracurium (Other): Patients who underwent general anesthesia received atracurium
  Interventions: Drug: atracurium
- cisatracurium (Other): Patients who underwent general anesthesia received cisatracurium
  Interventions: Drug: cisatracurium

INTERVENTIONS:
Drug: atracurium — atracurium, Drop,0.5 mg/kg, one time, one day
  Arms: atracurium
Drug: cisatracurium — cisatracurium, drop,0.15mg/kg,one time, one day
  Arms: cisatracurium

SUMMARY:
The purpose of this study is to determine which drug makes lower intraocular pressure

DETAILED DESCRIPTION:
Increase in intraocular pressure (IOP) following tracheal intubation during general anesthesia can be troublesome. The investigators compared the influence of cisatracurium and atracurium on IOP in patients undergoing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

ASA class of I or II baseline IOP of lower than 20 mmHg stable hemodynamics no history of ophthalmic diseases not using drugs affecting IOP (e.g. anticholinergics, sympathomimetics) no contraindication for atracurium or cisatracurium administration.

Exclusion Criteria:

difficulty in mask ventilation or in tracheal intubation end expiratory CO2 of below 35 mmHg or over 45 mmHg O2 saturation of below 90%

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
intraocular pressure | at 2 minutes after intubation
  determining intraocular pressure in atracurium and cisatracurium groups

SECONDARY OUTCOMES:
systolic blood pressure | at 2 minutes after intubation
  identification of systolic blood pressure in atracurium and cisatracurium groups

CONTACTS AND LOCATIONS:
Overall Officials: Mitra Jabalameri, A.Professor, Study Chair — Associate Professor,Anesthesiology department
Locations (1):
- Al-zahra university hospital, Isfahan, Isfahan, Iran